CLINICAL TRIAL: NCT05204355
Title: MRI for Screening and Monitoring Systemic Sclerosis Interstitial Lung Disease
Brief Title: MRI for Screening and Monitoring Scleroderma ILD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Scleroderma Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00148159
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scleroderma: Patients with Scleroderma will be imaged with UTE MRI to compare MRI with CT for identifying Interstitial Lung Disease
  Interventions: Diagnostic Test: MRI; Diagnostic Test: HRCT
- Scleroderma ILD: Patients with Scleroderma ILD who are initiating treatment will be imaged using hyperpolarized 129Xe MRI to assess treatment efficacy.
  Interventions: Diagnostic Test: MRI; Drug: Hyperpolarized Xe129

INTERVENTIONS:
Diagnostic Test: MRI — Patients will be imaged using MRI
Drug: Hyperpolarized Xe129 — Hyperpolarized Xe129 will be used to image the lungs of a subset of participants.
  Groups: Scleroderma ILD
Diagnostic Test: HRCT — High Resolution Computer Tomography
  Groups: Scleroderma

SUMMARY:
The purpose of this study is to test MRI methods for evaluating patients with Scleroderma-associated interstitial lung disease.

DETAILED DESCRIPTION:
1. Quantify the sensitivity and specificity of UTE MRI in screening for scleroderma-associated interstitial lung disease. ILD is relatively common in SSc, but current clinical standards require screening using HRCT. UTE MRI can provide images of pulmonary structure with contrast and resolution approaching that of CT. We hypothesize that UTE MRI will have high sensitivity and specificity (>80%) to the presence of ILD as determined by HRCT.

   Aim
2. Quantify treatment response in patients with SSc-ILD using hyperpolarized 129Xe MRI. The optimal treatment for SSc-ILD is not known, and it is challenging to assess the efficacy of therapy. Hyperpolarized 129Xe MRI is highly sensitive to the pathophysiology associated with ILD, which suggests that it may be more sensitive to treatment response than conventional methods. We hypothesize that hyperpolarized 129Xe MRI biomarkers will be sensitive to lung function improvement or decline earlier than standard clinical measures (6MWD, FVC, DLCO, Dyspnea score).

ELIGIBILITY:
Arm 1 (UTE MRI in patients with Scleroderma)

Inclusion Criteria:

* Age ≥ 18 years of age
* Subject has clinical diagnosis of scleroderma.
* Chest CT scan within 1 month prior to screening or Chest CT scan will be completed within 1 month post study enrollment.
* Ability to adhere to the study visit schedule, adhere, and comply with all protocol requirements.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Subject unable to undergo MRI based on MRI safety screening
* Pregnant or breastfeeding female subjects
* Prisoners or incarcerated individuals
* Any in-patient hospitalization (defined as greater than 23 hours) within 30 days of study enrollment
* Any major surgical procedure within 90 days prior to study enrollment or planned surgical procedure during the study period.
* Concomitant medical disorder, condition, or history, that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent or would confound the objectives of the study

Arm 2 (Hyperpolarized 129Xe MRI in Patients with Scleroderma ILD)

Inclusion Criteria:

* Age ≥ 18 years of age
* Subject clinically diagnosed with SSc-ILD.
* Subject initiating background SSc-ILD therapy within ±30 days of visit 1. (i.e. patient cannot have begun therapy for SSc-ILD more than 30 days prior to visit 1, or must be clinically scheduled to initiate therapy within 30 days after visit 1).
* FVC % Predicted ≥45% pre-bronchodilator within 30 days prior to screening or at baseline.
* DLCO % Predicted ≥30% within 30 days prior to screening or at baseline.
* Oxygen saturation >87% on room air or with supplemental oxygen
* Ability to adhere to the study visit schedule, adhere, and comply with all protocol requirements.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Subject unable to undergo MRI based on MRI safety screening
* Diagnosis of IPF based on ATS/ERS/JRS/ALAT 2018 Guidelines
* Significant Pulmonary Arterial Hypertension (PAH) defined by any of the following:

  1. Previous clinical or echocardiographic evidence of significant right heart failure
  2. History of right heart catheterization showing a cardiac index ≤ 2 l/min/m²
  3. PAH requiring parenteral therapy with epoprostenol/treprostinil
* Primary obstructive airway physiology (pre-bronchodilator FEV1/FVC < 0.7 at Baseline).
* Pregnant or breastfeeding female subjects
* Prisoners or incarcerated individuals
* Any in-patient hospitalization (defined as greater than 23 hours) within 30 days of study enrollment
* Any major surgical procedure within 90 days prior to study enrollment or planned surgical procedure during the study period.
* Concomitant medical disorder, condition, or history, that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent or would confound the objectives of the study
* Subject has been on therapy for SSc-ILD for >30 days prior to baseline MRI.
* Pregnancy (Visit 1 or Visit 2) or intention to become pregnant (Visit 2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be enrolled will have Scleroderma. Patients will be enrolled in either or both of arms 1 and 2:
  Arm 1: Patients with scleroderma who undergo a clinical CT scan to screen for ILD.
  Arm 2: Patients with scleroderma ILD who are initiating treatment for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Presence of ILD on CT and MRI | Baseline
  An experienced radiologist will review MRI and CT images to assess whether ILD is present.
Change in RBC/Barrier Ratio | 6 months
  The change in hyperpolarized 129Xe RBC/Barrier ratio from baseline to follow-up imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No